CLINICAL TRIAL: NCT06206577
Title: Autogenous Inlay Versus Onlay Grafts for Anterior Maxillary Horizontal Ridge Augmentation
Brief Title: Autogenous Grafts for Anterior Maxillary Horizontal Ridge Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Etman Elsayed, assisstant lecturer of oral and maxillofacial surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A08040820
Record Dates: First submitted 2023-12-20; First posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Alveolar Ridge Augmentation
Keywords: onlay grafting; inlay grafting

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Seven horizontal anterior maxillary ridge augmentation was done with symphyseal autogenous bone block, which was placed buccally as onlay graft.
  Interventions: Procedure: Horizontal ridge augmentation by symphyseal bone block placed and fixed buccally as onlay graft
- Group B (Experimental): Seven horizontal anterior maxillary ridge augmentation was done with symphyseal autogenous bone block, which was interpositioned in space created between buccal and lingual cortex as inlay graft.
  Interventions: Procedure: Horizontal ridge augmentation by symphyseal bone block interpositioned in space created between buccal and lingual cortex as inlay graft

INTERVENTIONS:
Procedure: Horizontal ridge augmentation by symphyseal bone block placed and fixed buccally as onlay graft — autogenous bone block harvested from chin area using piezosurgery and fixed buccally in deficient area with fixation screws
  Arms: Group A
Procedure: Horizontal ridge augmentation by symphyseal bone block interpositioned in space created between buccal and lingual cortex as inlay graft — autogenous bone block harvested from chin area using piezosurgery and fixed in bone split created at deficient area with fixation screws
  Arms: Group B

SUMMARY:
The aim of the study was to compare efficacy of autogenous onlay and inlay grafts for anterior maxillary horizontal ridge augmentation.

DETAILED DESCRIPTION:
Autogenous block graft has been used as onlay thin cortical shell and cortico-cancellous particles. The thin cortical shell acts as an autogenous biological membrane that will resist resorption and stabilize the small pieces of particulate bone. The bone block is screwed-in at a distance from the recipient site by means of titanium bone screws, and then the free space under the shell is filled with the particulate bone.

The resultant augmentation somehow resembles an iliac graft, with thick internal cancellous bone and a thin external cortical layer. This leads to an ideal graft, with a high regenerative capacity comparable to iliac bone and a stable regenerated volume with optimum osseointegration potential close to that of mandibular block grafts.

Interpositional grafts have been successfully established in restoring vertical bone height . However much less evidence is present on its use for horizontal augmentation. It is the purpose of this study to assess the efficacy of autogenous onlay corticocancellous block grafts for anterior maxillary horizontal ridge augmentation as compared to onlay block grafts.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with missing upper anterior tooth / teeth with horizontal ridge dimension range from 2 to 5 mm (measured 2mm below alveolar crest).
2. Adequate vertical height.
3. Having good oral hygiene.
4. being healthy, with no systemic diseases that might contraindicate receiving a dental implant
5. Patients were able to comply with the follow-up and maintenance program

Exclusion Criteria:

1. Presence of local infection or lesions at site of interest.
2. Dental history of bruxism, or other parafunctional habits.
3. Uncooperative patients.
4. Current chemotherapy or radiotherapy.
5. Patients with aggressive periodontal disease

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
horizontal ridge augmentation | 12 months
  CBCT to assess bone gain in mm

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura U, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No